CLINICAL TRIAL: NCT00461474
Title: Strengthening and Optimal Movements for Painful Shoulders in Chronic Spinal Cord Injury (STOMPS)
Brief Title: Study of Strengthening Exercises and Improving Movement for Painful Shoulders in Adults With Spinal Cord Injury
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: Physical Therapy Clinical Research Network (Network)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HS-025022
Record Dates: First submitted 2007-04-16; First posted 2007-04-18 (Estimated); Last update posted 2007-04-19 (Estimated); Status verified 2007-04

CONDITIONS: Shoulder Pain
Keywords: Shoulder pain; Chronic Spinal Cord Injury; Exercise; Physical therapy techniques; Motor performance
MeSH Terms: conditions — Shoulder Pain; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Shoulder strengthening exercises
Behavioral: Movement Optimization

SUMMARY:
The purpose of this study is to conduct research to see if we can help people who have a spinal cord injury and shoulder pain to decrease the pain in the shoulders. We are investigating the effectiveness of a home exercise program for the shoulders and changes in how tasks are performed compared to an educational program on shoulder pain. There are no new experimental procedures included in this study; instead it is a comparison of two types of treatment that have been provided for this problem before. The new part of this study is the collecting of information before and after treatment. We hypothesize that those who participate in this home exercise program will have decrease shoulder pain and increase activity.

DETAILED DESCRIPTION:
Adults who sustain a spinal cord injury (SCI) now have the potential to lead active, productive lives with near normal life expectancy. Recent studies have demonstrated that many people with SCI develop health and functional problems at earlier ages than their non-disabled peers, with symptoms often occurring between the mid-30's and the mid-50's. These symptoms and impairments include: pain, musculoskeletal problems, declining energy, loss of strength and new functional limitations. These are examples of the challenges people may face as they reach mid-life with a SCI. A prevalent impairment in the long-term SCI population is upper extremity pain. Both the incidence and severity of pain increase with longer duration of SCI. The impact of shoulder pain on function and independence after SCI can be significant and detrimental. Development of shoulder pain in the SCI population has been associated with the increased weight-bearing demand placed on the upper extremities for mobility, muscle imbalances in the shoulder girdle, poor postural alignment from trunk paralysis and the need to function from a seated position. The efficacy of specific interventions has not been fully investigated. Treatment effectiveness must be determined using measures that include the pain impairment (severity), the disability or functional limitation associated with pain, and the participation or handicap limitations associated with pain. The goal is to develop a program that has standardized resistance, requires little equipment, is simple to conduct and minimizes the time commitment required of the patient. The effect of the combined intervention on shoulder pain and function will be assessed with a randomized clinical trial comparing the intervention to an attention control group receiving generalized information regarding shoulder joint anatomy and pain management. Secondary goals of this study are to identify the critical muscle groups for which strength changes are associated with shoulder pain reduction and to determine the impact of the intervention on physical activity, health related quality of life and overall subjective quality of life.

ELIGIBILITY:
Inclusion Criteria:

* post-pubescent (age 14 or older) onset of paraplegia,
* at least 5 years duration with spinal cord injury, current age between 19 and 75,
* unilateral or bilateral shoulder pain that interferes with at least one functional task (e.g. transfers, wheelchair propulsion),
* subjects who propel a manual wheelchair >50% normalized velocity and ability to understand the informed consent.

Exclusion Criteria:

* hospitalization within the last month
* a cortisone injection to the shoulder within the last 4 months,
* a fracture within the last year,
* shoulder surgery to the painful side within the last year,
* a diagnosis of complete rotator cuff tear, rheumatoid arthritis, adhesive capsulitis at the shoulder or complex regional pain syndrome (also known as reflex sympathetic dystrophy),
* any serious medical conditions, major depression, alcohol abuse, or being unlikely to complete the 12-weeks of treatment.

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80
Dates: Start 2004-03; Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
shoulder pain as measured by Wheelchair Users Shoulder Pain Index (WUSPI)

SECONDARY OUTCOMES:
General shoulder pain measured by a visual analog scale (VAS)from the McGill Short Form Pain Questionnaire
Shoulder torque with a hand held dynamometer
Subject's activity level with the Physical Activity Scale for Individuals with Physical Disabilities (PASIPD)
Community involvement with the Community Activities Checklist (CAC)
Quality of life with the SF-36 Health Related Quality of Life questionnaire
Quality of life with the Subjective Quality of Life Scale (SQOL)
Wheelchair propulsion

CONTACTS AND LOCATIONS:
Overall Officials: Bryan Kemp, Ph.D, Principal Investigator — Rancho Los Amigos National Rehabilitation Center; Carolee J. Winstein, Ph.D., PT, Principal Investigator — University of Southern California; Sara Mulroy, Ph.D., PT, Principal Investigator — Rancho Los Amigos National Rehabilitation Center
Locations (1):
- Rancho Los Amigos National Rehabilitation Hospital, Downey, California, United States